CLINICAL TRIAL: NCT00938015
Title: A Post-Marketing Surveillance For Safety And Adherence To Treatment Of Enbrel In Adults With Psoriatic Arthritis In Belgium
Brief Title: Study Evaluating Safety and Adherence to Treatment With Etanercept in Adults With Psoriatic Arthritis
Acronym: PROVE
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: 0881A-101698; B1801107
Record Dates: First submitted 2009-07-10; First posted 2009-07-13 (Estimated); Results first posted 2013-05-27 (Estimated); Last update posted 2013-05-27 (Estimated); Status verified 2013-03

CONDITIONS: Arthritis, Psoriatic
Keywords: postmarketing surveillance; Enbrel; psoriatic arthritis
MeSH Terms: conditions — Arthritis, Psoriatic | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- PsA Patients (New): New patients
  Interventions: Other: Questionnaire
- PsA Patients: CU patients
  Interventions: Other: Questionnaire

INTERVENTIONS:
Other: Questionnaire — This is a non-interventional study
  Groups: PsA Patients (New)
Other: Questionnaire — This is a non-interventional study
  Groups: PsA Patients

SUMMARY:
The aim of this study is to evaluate if the data obtained in controlled clinical trials are confirmed when Enbrel is used in usual clinical practice in Belgium according to local reimbursement criteria.

ELIGIBILITY:
Inclusion Criteria:

* Active erosive psoriatic arthritis of poly-articular type or active erosive or with joint space narrowing psoriatic arthritis of oligo-articular type
* At least 18 years old
* Have fulfilled reimbursement criteria for Enbrel in psoriatic arthritis of poly-articular type or oligo-articular type
* Physician decides to prescribe Enbrel or patient is already on Enbrel
* Give written informed consent at time of inclusion to study

Exclusion Criteria:

NA

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: rheumatology centers
Sampling Method: Non-Probability Sample
Enrollment: 303 (Actual)
Dates: Start 2004-10; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, Leuven, Belgium

REFERENCES:
- [Derived] de Vlam K, Boone C, The Prove Study Group A. Treatment adherence, efficacy, and safety of etanercept in patients with active psoriatic arthritis and peripheral involvement in Belgium for 66 months (PROVE study). Clin Exp Rheumatol. 2015 Sep-Oct;33(5):624-31. Epub 2015 Jul 23. PMID 26212872
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=0881A-101698&StudyName=Study%20Evaluating%20Safety%20and%20Adherence%20to%20Treatment%20with%20Etanercept%20in%20Adults%20with%20Psoriatic%20Arthritis

RESULTS

PARTICIPANT FLOW:
Groups:
- Etanercept: Participants with psoriatic arthritis (PsA) who received etanercept (Enbrel) as per standard practice were observed for 6.5 years.
Period: Overall Study
Arm/Group | Etanercept
Started | 303
Completed | 156
Not Completed | 147
Not completed — Death | 2
Not completed — Lost to Follow-up | 32
Not completed — Adverse Event | 32
Not completed — Non-responder | 52
Not completed — Reason not related to Etanercept | 29

BASELINE CHARACTERISTICS:
Arm/Group | Etanercept
Number analyzed (Participants) | 303
Age Continuous [Mean (Standard Deviation); unit: Years] | 48.29 (10.83)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 137
  Male | 166

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With at Least 1 Serious Adverse Event (SAE): Baseline up to Year 1
Description: An adverse event (AE) was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. An SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly.
Time Frame: Baseline up to Year 1
Population: Safety set included all the participants who signed informed consent form (ICF) and had at least one dose of study medication and had follow-up data.
Measure: Number; unit: Percentage of participants
Arm/Group | Etanercept
Number analyzed (Participants) | 301
Percentage of participants | 7.97

2. Primary Outcome: Percentage of Participants With at Least 1 Serious Adverse Event (SAE): Year 1 up to Year 2
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. An SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly.
Time Frame: Year 1 up to Year 2
Population: Safety set included all the participants who signed ICF and had at least one dose of study medication and had follow-up data. 'N' (number of participants analyzed) signifies those participants who were evaluable for this measure.
Measure: Number; unit: Percentage of participants
Arm/Group | Etanercept
Number analyzed (Participants) | 278
Percentage of participants | 7.91

3. Primary Outcome: Percentage of Participants With at Least 1 Serious Adverse Event (SAE): Year 2 up to Year 3
Description: as for outcome 2
Time Frame: Year 2 up to Year 3
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | Etanercept
Number analyzed (Participants) | 227
Percentage of participants | 4.85

4. Primary Outcome: Percentage of Participants With at Least 1 Serious Adverse Event (SAE): Year 3 up to Year 4
Description: as for outcome 2
Time Frame: Year 3 up to Year 4
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | Etanercept
Number analyzed (Participants) | 198
Percentage of participants | 4.55

5. Primary Outcome: Percentage of Participants With at Least 1 Serious Adverse Event (SAE): Year 4 up to Year 5
Description: as for outcome 2
Time Frame: Year 4 up to Year 5
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | Etanercept
Number analyzed (Participants) | 178
Percentage of participants | 3.37

6. Primary Outcome: Percentage of Participants With at Least 1 Serious Adverse Event (SAE): Year 5 up to Year 6
Description: as for outcome 2
Time Frame: Year 5 up to Year 6
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | Etanercept
Number analyzed (Participants) | 159
Percentage of participants | 2.52

7. Secondary Outcome: Percentage of Participants With at Least 1 Adverse Event (AE) Per Year
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship.
Time Frame: Baseline up to Year 6
Population: Safety set included all the participants who signed ICF and had at least one dose of study medication and had follow-up data. 'n' signifies those participants who were evaluable for this measure at given time points.
Measure: Number; unit: Percentage of participants
Arm/Group | Etanercept
Number analyzed (Participants) | 301
Percentage of participants
  Till Year 1 (n=301) | 44.19
  Year 1 to Year 2 (n=278) | 37.77
  Year 2 to Year 3 (n=227) | 33.92
  Year 3 to Year 4 (n=198) | 34.85
  Year 4 to Year 5 (n=178) | 31.46
  Year 5 to Year 6 (n=159) | 21.38

8. Secondary Outcome: Incidence of Adverse Events and Serious Adverse Events Per Participant-Year
Description: Participant-Year estimated by calculating all of the years that participants in a study were followed (mean study drug exposure duration multiplied by safety set population). Incidence calculated as AEs or SAEs divided by Participant-Year multiplied by 100. Incidence of AEs and SAEs were broken down by each follow-up time period.
Time Frame: Baseline up to Month 6, 12, 18, 30, 42, 54, 66
Population: as for outcome 7
Measure: Number; unit: Events per participant year
Arm/Group | Etanercept
Number analyzed (Participants) | 301
Events per participant year
  Incidence of AEs till Month 6 | 145.68
  Incidence of AEs till Month 12 | 138.51
  Incidence of AEs till Month 18 | 134.23
  Incidence of AEs till Month 30 | 125.73
  Incidence of AEs till Month 42 | 117.93
  Incidence of AEs till Month 54 | 118.49
  Incidence of AEs till Month 66 | 112.79
  Incidence of SAEs till Month 6 | 9.44
  Incidence of SAEs till Month 12 | 14.54
  Incidence of SAEs till Month 18 | 13.23
  Incidence of SAEs till Month 30 | 14.11
  Incidence of SAEs till Month 42 | 12.23
  Incidence of SAEs till Month 54 | 11.29
  Incidence of SAEs till Month 66 | 10.65

9. Secondary Outcome: Percentage of Participants With Psoriatic Arthritis (PsA) Receiving Enbrel Who Stayed on the Treatment
Time Frame: Baseline up to Month 78
Population: Efficacy set included all the participants who signed ICF.
Measure: Number; unit: Percentage of participants
Arm/Group | Etanercept
Number analyzed (Participants) | 303
Percentage of participants | 51.49

10. Secondary Outcome: Number of Joints With Active Arthritis
Description: Numbers of joints with active arthritis were defined as joints that were swollen or, in absence of swelling, joints with limited motion with pain and/or tenderness.
Time Frame: Baseline, Month 6, Month 12, Month 18, Month 30, Month 42, Month 54, Month 66, Month 78
Population: Efficacy set included all the participants who signed ICF. 'N' (Number of participants analyzed) signifies those participants who were evaluable for this measure and 'n' signifies those participants who were evaluable for this measure at given time points.
Measure: Mean (Standard Deviation); unit: Joints
Arm/Group | Etanercept
Number analyzed (Participants) | 302
Joints
  Baseline (n=302) | 11.81 (6.77)
  Month 6 (n=288) | 2.10 (3.36)
  Month 12 (n=260) | 1.80 (4.65)
  Month 18 (n=261) | 1.34 (3.45)
  Month 30 (n=215) | 1.13 (2.91)
  Month 42 (n=189) | 0.83 (2.17)
  Month 54 (n=169) | 0.77 (2.47)
  Month 66 (n=152) | 0.73 (2.00)
  Month 78 (n=5) | 1.00 (1.41)

11. Secondary Outcome: Quality of Life Assessed by Numerical Rating Scale (NRS) For Oligo-Articular Type Psoriatic Arthritis (PsA) - Participant Evaluation
Description: Quality of life for oligo-articular type arthritis was assessed on a 11-point Numerical Rating Scale (NRS) ranging from 1 (best health status) to 10 (worst health status). NRS for the most affected joint as per participant was evaluated.
Time Frame: Baseline, Month 6, Month 12, Month 18, Month 30, Month 42, Month 54, Month 66, Month 78
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Etanercept
Number analyzed (Participants) | 37
Units on a scale
  Baseline (n=37) | 7.35 (1.46)
  Month 6 (n=27) | 3.33 (1.84)
  Month 12 (n=19) | 3.16 (1.83)
  Month 18 (n=24) | 3.29 (2.42)
  Month 30 (n=18) | 3.00 (1.64)
  Month 42 (n=13) | 2.23 (1.42)
  Month 54 (n=9) | 3.11 (2.57)
  Month 66 (n=5) | 3.80 (3.03)
  Month 78 (n=0) | NA (NA) — Data was not analyzed as there was no participant evaluable for this category at given time point.

12. Secondary Outcome: Quality of Life Assessed by Numerical Rating Scale (NRS) For Oligo-Articular Type Psoriatic Arthritis (PsA) - Physician Evaluation
Description: Quality of life for oligo-articular type arthritis was assessed on a 11-point NRS ranging from 1 (best health status) to 10 (worst health status). NRS for the most affected joint as per physician was evaluated.
Time Frame: Baseline, Month 6, Month 12, Month 18, Month 30, Month 42, Month 54, Month 66, Month 78
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Etanercept
Number analyzed (Participants) | 37
Units on a scale
  Baseline (n=37) | 6.51 (1.22)
  Month 6 (n=27) | 2.44 (1.48)
  Month 12 (n=20) | 2.35 (1.35)
  Month 18 (n=24) | 2.50 (1.96)
  Month 30 (n=18) | 2.22 (1.11)
  Month 42 (n=13) | 1.77 (0.73)
  Month 54 (n=9) | 2.11 (1.45)
  Month 66 (n=5) | 3.40 (2.79)
  Month 78 (n=0) | NA (NA) — Data was not analyzed as there was no participant evaluable for this category at given time point.

13. Secondary Outcome: Quality of Life Assessed by Health Assessment Questionnaire (HAQ) For Poly-Articular Type Psoriatic Arthritis (PsA)
Description: HAQ is a 20 item questionnaire to measure functional limitations. Participants were rated on 4 point scale with scores: 0=no difficulty (normal), 1=some difficulty (adequate), 2=much difficulty (limited), 3=unable to do based on degree of difficulty experienced with 20 items grouped into 8 areas of dressing, rising, hygiene, reach, walking, eating, grip and activities. Total score range 0-60, higher score indicating greater functional limitations.
Time Frame: Baseline, Month 6, Month 12, Month 18, Month 30, Month 42, Month 54, Month 66, Month 78
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Etanercept
Number analyzed (Participants) | 261
Units on a scale
  Baseline (n=261) | 26.99 (8.94)
  Month 6 (n=239) | 9.72 (9.37)
  Month 12 (n=194) | 8.87 (9.51)
  Month 18 (n=209) | 8.09 (9.20)
  Month 30 (n=182) | 7.75 (8.93)
  Month 42 (n=166) | 7.16 (8.63)
  Month 54 (n=149) | 7.43 (8.40)
  Month 66 (n=135) | 7.70 (9.09)
  Month 78 (n=4) | 15.75 (10.31)

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | Etanercept
Serious Adverse Events (participants affected / at risk) | 65/301
Other Adverse Events (participants affected / at risk) | 179/301
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Etanercept (N=301)
Acute myocardial infarction (Cardiac disorders) | 2
Angina pectoris (Cardiac disorders) | 1
Atrial fibrillation (Cardiac disorders) | 3
Coronary artery disease (Cardiac disorders) | 1
Vertigo (Ear and labyrinth disorders) | 1
Vestibular neuronitis (Ear and labyrinth disorders) | 1
Corneal erosion (Eye disorders) | 1
Diplopia (Eye disorders) | 1
Abdominal pain lower (Gastrointestinal disorders) | 1
Colitis ulcerative (Gastrointestinal disorders) | 1
Colonic polyp (Gastrointestinal disorders) | 1
Crohn's disease (Gastrointestinal disorders) | 1
Pancreatitis (Gastrointestinal disorders) | 1
Pancreatitis acute (Gastrointestinal disorders) | 1
Condition aggravated (General disorders) | 3
Fatigue (General disorders) | 1
Cholecystitis acute (Hepatobiliary disorders) | 1
Hepatic failure (Hepatobiliary disorders) | 1
Hepatic steatosis (Hepatobiliary disorders) | 1
Arthritis bacterial (Infections and infestations) | 1
Cellulitis (Infections and infestations) | 2
Escherichia sepsis (Infections and infestations) | 1
Hepatitis C (Infections and infestations) | 1
Herpes zoster ophthalmic (Infections and infestations) | 1
Keratitis herpetic (Infections and infestations) | 1
Localised infection (Infections and infestations) | 1
Osteomyelitis (Infections and infestations) | 1
Otitis media (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 2
Prostatic abscess (Infections and infestations) | 1
Respiratory tract infection (Infections and infestations) | 1
Septic shock (Infections and infestations) | 1
Staphylococcal bacteraemia (Infections and infestations) | 1
Urosepsis (Infections and infestations) | 1
Femoral neck fracture (Injury, poisoning and procedural complications) | 1
Ligament rupture (Injury, poisoning and procedural complications) | 1
Rib fracture (Injury, poisoning and procedural complications) | 1
Scapula fracture (Injury, poisoning and procedural complications) | 1
Splenic rupture (Injury, poisoning and procedural complications) | 1
Subdural haematoma (Injury, poisoning and procedural complications) | 1
Tendon rupture (Injury, poisoning and procedural complications) | 3
Hepatic enzyme increased (Investigations) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 2
Back pain (Musculoskeletal and connective tissue disorders) | 2
Bone cyst (Musculoskeletal and connective tissue disorders) | 1
Bursitis (Musculoskeletal and connective tissue disorders) | 2
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1
Joint destruction (Musculoskeletal and connective tissue disorders) | 1
Psoriatic arthropathy (Musculoskeletal and connective tissue disorders) | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Lung adenocarcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Amnestic disorder (Nervous system disorders) | 1
Cerebrovascular accident (Nervous system disorders) | 1
Cognitive disorder (Nervous system disorders) | 1
Demyelination (Nervous system disorders) | 1
Headache (Nervous system disorders) | 1
Multiple sclerosis (Nervous system disorders) | 1
Depression (Psychiatric disorders) | 2
Nephrolithiasis (Renal and urinary disorders) | 1
Renal colic (Renal and urinary disorders) | 1
Renal impairment (Renal and urinary disorders) | 1
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1
Alveolitis allergic (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 2
Arthrodesis (Surgical and medical procedures) | 1
Bladder operation (Surgical and medical procedures) | 1
Bunion operation (Surgical and medical procedures) | 1
Cataract operation (Surgical and medical procedures) | 1
Cholecystectomy (Surgical and medical procedures) | 1
Chondroplasty (Surgical and medical procedures) | 1
Hernia repair (Surgical and medical procedures) | 1
Internal fixation of fracture (Surgical and medical procedures) | 1
Knee arthroplasty (Surgical and medical procedures) | 1
Prostatic operation (Surgical and medical procedures) | 1
Sinus operation (Surgical and medical procedures) | 1
Synovectomy (Surgical and medical procedures) | 2
Toe operation (Surgical and medical procedures) | 1
Varicose vein operation (Surgical and medical procedures) | 1
Deep vein thrombosis (Vascular disorders) | 2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Etanercept (N=301)
Anaemia (Blood and lymphatic system disorders) | 1
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1
Leukopenia (Blood and lymphatic system disorders) | 7
Lymphadenitis (Blood and lymphatic system disorders) | 1
Lymphadenopathy (Blood and lymphatic system disorders) | 2
Macrocytosis (Blood and lymphatic system disorders) | 1
Neutropenia (Blood and lymphatic system disorders) | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 1
Atrial fibrillation (Cardiac disorders) | 1
Bradycardia (Cardiac disorders) | 1
Palpitations (Cardiac disorders) | 6
Tachycardia (Cardiac disorders) | 3
Ear pain (Ear and labyrinth disorders) | 2
Vertigo (Ear and labyrinth disorders) | 3
Hyperthyroidism (Endocrine disorders) | 1
Hypothyroidism (Endocrine disorders) | 1
Conjunctival hyperaemia (Eye disorders) | 1
Conjunctivitis (Eye disorders) | 5
Dry eye (Eye disorders) | 4
Eye irritation (Eye disorders) | 3
Eye pruritus (Eye disorders) | 2
Glaucoma (Eye disorders) | 1
Lacrimation increased (Eye disorders) | 1
Uveitis (Eye disorders) | 2
Visual acuity reduced (Eye disorders) | 1
Visual disturbance (Eye disorders) | 2
Abdominal discomfort (Gastrointestinal disorders) | 2
Abdominal pain (Gastrointestinal disorders) | 1
Abdominal pain upper (Gastrointestinal disorders) | 8
Aphthous stomatitis (Gastrointestinal disorders) | 1
Colitis (Gastrointestinal disorders) | 1
Colonic polyp (Gastrointestinal disorders) | 2
Constipation (Gastrointestinal disorders) | 1
Crohn's disease (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 16
Dry mouth (Gastrointestinal disorders) | 1
Dyspepsia (Gastrointestinal disorders) | 5
Enteritis (Gastrointestinal disorders) | 1
Epiploic appendagitis (Gastrointestinal disorders) | 1
Frequent bowel movements (Gastrointestinal disorders) | 1
Gastric ulcer (Gastrointestinal disorders) | 3
Gastritis (Gastrointestinal disorders) | 1
Gastrointestinal disorder (Gastrointestinal disorders) | 1
Gastrointestinal pain (Gastrointestinal disorders) | 1
Gastrooesophagitis (Gastrointestinal disorders) | 1
Gingivitis (Gastrointestinal disorders) | 2
Haemorrhoids (Gastrointestinal disorders) | 2
Hiatus hernia (Gastrointestinal disorders) | 1
Inguinal hernia (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 10
Pancreatitis (Gastrointestinal disorders) | 1
Periodontitis (Gastrointestinal disorders) | 1
Reflux oesophagitis (Gastrointestinal disorders) | 4
Stomach discomfort (Gastrointestinal disorders) | 1
Toothache (Gastrointestinal disorders) | 3
Vomiting (Gastrointestinal disorders) | 3
Asthenia (General disorders) | 2
Chest pain (General disorders) | 1
Chills (General disorders) | 1
Drug intolerance (General disorders) | 1
Fatigue (General disorders) | 18
Haemorrhagic cyst (General disorders) | 1
Impaired healing (General disorders) | 2
Influenza like illness (General disorders) | 9
Injection site erythema (General disorders) | 1
Injection site irritation (General disorders) | 1
Injection site pruritus (General disorders) | 1
Injection site rash (General disorders) | 2
Injection site reaction (General disorders) | 1
Malaise (General disorders) | 1
Pyrexia (General disorders) | 11
Rebound effect (General disorders) | 1
Cholelithiasis (Hepatobiliary disorders) | 1
Cirrhosis alcoholic (Hepatobiliary disorders) | 1
Hepatic function abnormal (Hepatobiliary disorders) | 15
Hepatic steatosis (Hepatobiliary disorders) | 4
Allergy to arthropod sting (Immune system disorders) | 1
Atopy (Immune system disorders) | 1
Hypersensitivity (Immune system disorders) | 2
Seasonal allergy (Immune system disorders) | 1
Acute tonsillitis (Infections and infestations) | 7
Anogenital warts (Infections and infestations) | 1
Bronchitis (Infections and infestations) | 17
Cystitis (Infections and infestations) | 3
Cystitis escherichia (Infections and infestations) | 1
Ear infection (Infections and infestations) | 2
Epiglottitis (Infections and infestations) | 1
Erysipelas (Infections and infestations) | 2
Eye infection (Infections and infestations) | 3
Folliculitis (Infections and infestations) | 1
Fungal infection (Infections and infestations) | 1
Furuncle (Infections and infestations) | 1
Gastroenteritis (Infections and infestations) | 7
Gastrointestinal fungal infection (Infections and infestations) | 1
Gastrointestinal infection (Infections and infestations) | 1
Genital infection male (Infections and infestations) | 1
Helicobacter gastritis (Infections and infestations) | 2
Herpes simplex (Infections and infestations) | 5
Herpes zoster (Infections and infestations) | 5
Infection (Infections and infestations) | 1
Influenza (Infections and infestations) | 15
Laryngitis (Infections and infestations) | 2
Molluscum contagiosum (Infections and infestations) | 1
Nail infection (Infections and infestations) | 1
Nasopharyngitis (Infections and infestations) | 41
Onychomycosis (Infections and infestations) | 1
Oral fungal infection (Infections and infestations) | 1
Orchitis (Infections and infestations) | 1
Otitis externa (Infections and infestations) | 1
Otitis media (Infections and infestations) | 2
Parotitis (Infections and infestations) | 1
Pharyngitis (Infections and infestations) | 4
Pneumonia (Infections and infestations) | 1
Pneumonia mycoplasmal (Infections and infestations) | 1
Respiratory tract infection (Infections and infestations) | 4
Respiratory tract infection fungal (Infections and infestations) | 1
Respiratory tract infection viral (Infections and infestations) | 1
Rhinitis (Infections and infestations) | 4
Sinusitis (Infections and infestations) | 17
Skin infection (Infections and infestations) | 1
Staphylococcal infection (Infections and infestations) | 1
Subcutaneous abscess (Infections and infestations) | 1
Tinea versicolour (Infections and infestations) | 2
Tooth abscess (Infections and infestations) | 1
Tooth infection (Infections and infestations) | 2
Tracheitis (Infections and infestations) | 1
Upper respiratory tract infection (Infections and infestations) | 24
Urethritis (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 8
Vaginal infection (Infections and infestations) | 1
Viral infection (Infections and infestations) | 1
Viral sinusitis (Infections and infestations) | 1
Wound infection (Infections and infestations) | 1
Accident at work (Injury, poisoning and procedural complications) | 1
Animal bite (Injury, poisoning and procedural complications) | 1
Arthropod bite (Injury, poisoning and procedural complications) | 1
Arthropod sting (Injury, poisoning and procedural complications) | 1
Contusion (Injury, poisoning and procedural complications) | 1
Epicondylitis (Injury, poisoning and procedural complications) | 4
Fall (Injury, poisoning and procedural complications) | 7
Foot fracture (Injury, poisoning and procedural complications) | 3
Foreign body in eye (Injury, poisoning and procedural complications) | 1
Fracture (Injury, poisoning and procedural complications) | 1
Heat stroke (Injury, poisoning and procedural complications) | 1
Impacted fracture (Injury, poisoning and procedural complications) | 1
Injury (Injury, poisoning and procedural complications) | 1
Joint sprain (Injury, poisoning and procedural complications) | 3
Meniscus lesion (Injury, poisoning and procedural complications) | 1
Muscle rupture (Injury, poisoning and procedural complications) | 1
Patella fracture (Injury, poisoning and procedural complications) | 1
Radius fracture (Injury, poisoning and procedural complications) | 1
Road traffic accident (Injury, poisoning and procedural complications) | 1
Synovial rupture (Injury, poisoning and procedural complications) | 1
Tendon rupture (Injury, poisoning and procedural complications) | 2
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 1
Tibia fracture (Injury, poisoning and procedural complications) | 1
Traumatic fracture (Injury, poisoning and procedural complications) | 1
Ulnar nerve injury (Injury, poisoning and procedural complications) | 1
Upper limb fracture (Injury, poisoning and procedural complications) | 1
Wound (Injury, poisoning and procedural complications) | 4
Wrist fracture (Injury, poisoning and procedural complications) | 1
Alanine aminotransferase increased (Investigations) | 2
Aspartate aminotransferase increased (Investigations) | 1
Blood cholesterol increased (Investigations) | 1
Blood creatine phosphokinase increased (Investigations) | 1
Blood glucose increased (Investigations) | 1
Blood triglycerides increased (Investigations) | 1
Gamma-glutamyltransferase increased (Investigations) | 2
Intraocular pressure increased (Investigations) | 1
Liver function test abnormal (Investigations) | 4
Monoclonal immunoglobulin present (Investigations) | 1
Transaminases increased (Investigations) | 3
Weight increased (Investigations) | 1
White blood cell count decreased (Investigations) | 1
Gout (Metabolism and nutrition disorders) | 1
Hypercholesterolaemia (Metabolism and nutrition disorders) | 2
Hyperglycaemia (Metabolism and nutrition disorders) | 1
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 1
Hypokalaemia (Metabolism and nutrition disorders) | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 3
Arthritis (Musculoskeletal and connective tissue disorders) | 1
Arthropathy (Musculoskeletal and connective tissue disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 8
Bursitis (Musculoskeletal and connective tissue disorders) | 7
Fibromyalgia (Musculoskeletal and connective tissue disorders) | 1
Gouty tophus (Musculoskeletal and connective tissue disorders) | 1
Groin pain (Musculoskeletal and connective tissue disorders) | 2
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 1
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 3
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1
Muscle rigidity (Musculoskeletal and connective tissue disorders) | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 3
Neck pain (Musculoskeletal and connective tissue disorders) | 2
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 4
Osteopenia (Musculoskeletal and connective tissue disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2
Periarthritis (Musculoskeletal and connective tissue disorders) | 1
Psoriatic arthropathy (Musculoskeletal and connective tissue disorders) | 4
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 3
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 2
Synovitis (Musculoskeletal and connective tissue disorders) | 1
Tendon disorder (Musculoskeletal and connective tissue disorders) | 1
Tendonitis (Musculoskeletal and connective tissue disorders) | 8
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 1
Adrenal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Balance disorder (Nervous system disorders) | 1
Carotid artery stenosis (Nervous system disorders) | 1
Carpal tunnel syndrome (Nervous system disorders) | 2
Disturbance in attention (Nervous system disorders) | 1
Dizziness (Nervous system disorders) | 3
Dizziness postural (Nervous system disorders) | 1
Headache (Nervous system disorders) | 17
Memory impairment (Nervous system disorders) | 1
Paraesthesia (Nervous system disorders) | 3
Sciatica (Nervous system disorders) | 1
Somnolence (Nervous system disorders) | 1
Syncope (Nervous system disorders) | 2
Syncope vasovagal (Nervous system disorders) | 1
Tremor (Nervous system disorders) | 2
Vertebral artery stenosis (Nervous system disorders) | 1
Alcoholism (Psychiatric disorders) | 1
Confusional state (Psychiatric disorders) | 1
Depressed mood (Psychiatric disorders) | 6
Depression (Psychiatric disorders) | 2
Insomnia (Psychiatric disorders) | 4
Nervousness (Psychiatric disorders) | 1
Obsessive-compulsive disorder (Psychiatric disorders) | 1
Stress (Psychiatric disorders) | 1
Calculus urinary (Renal and urinary disorders) | 2
Haematuria (Renal and urinary disorders) | 1
Micturition urgency (Renal and urinary disorders) | 1
Nephroangiosclerosis (Renal and urinary disorders) | 1
Nephrolithiasis (Renal and urinary disorders) | 4
Renal colic (Renal and urinary disorders) | 3
Renal impairment (Renal and urinary disorders) | 4
Urinary incontinence (Renal and urinary disorders) | 1
Balanitis (Reproductive system and breast disorders) | 1
Breast mass (Reproductive system and breast disorders) | 1
Epididymitis (Reproductive system and breast disorders) | 1
Erectile dysfunction (Reproductive system and breast disorders) | 3
Prostatitis (Reproductive system and breast disorders) | 1
Retracted nipple (Reproductive system and breast disorders) | 1
Uterine polyp (Reproductive system and breast disorders) | 1
Varicocele (Reproductive system and breast disorders) | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 19
Diaphragmatic hernia (Respiratory, thoracic and mediastinal disorders) | 1
Dry throat (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 2
Hyperventilation (Respiratory, thoracic and mediastinal disorders) | 2
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 1
Obliterative bronchiolitis (Respiratory, thoracic and mediastinal disorders) | 1
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 9
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 3
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1
Sneezing (Respiratory, thoracic and mediastinal disorders) | 1
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 1
Vasomotor rhinitis (Respiratory, thoracic and mediastinal disorders) | 1
Alopecia (Skin and subcutaneous tissue disorders) | 3
Blister (Skin and subcutaneous tissue disorders) | 1
Dermatitis (Skin and subcutaneous tissue disorders) | 1
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 4
Erythema (Skin and subcutaneous tissue disorders) | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 2
Neurodermatitis (Skin and subcutaneous tissue disorders) | 1
Night sweats (Skin and subcutaneous tissue disorders) | 2
Petechiae (Skin and subcutaneous tissue disorders) | 2
Pruritus (Skin and subcutaneous tissue disorders) | 3
Psoriasis (Skin and subcutaneous tissue disorders) | 10
Rash (Skin and subcutaneous tissue disorders) | 6
Rosacea (Skin and subcutaneous tissue disorders) | 1
Skin haemorrhage (Skin and subcutaneous tissue disorders) | 1
Skin lesion (Skin and subcutaneous tissue disorders) | 1
Toxic skin eruption (Skin and subcutaneous tissue disorders) | 1
Urticaria (Skin and subcutaneous tissue disorders) | 4
Tobacco abuse (Social circumstances) | 1
Colon polypectomy (Surgical and medical procedures) | 1
Finger repair operation (Surgical and medical procedures) | 1
Foot operation (Surgical and medical procedures) | 1
Gastric banding (Surgical and medical procedures) | 1
Knee arthroplasty (Surgical and medical procedures) | 1
Knee operation (Surgical and medical procedures) | 1
Meniscus removal (Surgical and medical procedures) | 1
Osteotomy (Surgical and medical procedures) | 1
Shoulder operation (Surgical and medical procedures) | 1
Sinus operation (Surgical and medical procedures) | 1
Skin lesion excision (Surgical and medical procedures) | 1
Toe operation (Surgical and medical procedures) | 1
Tooth extraction (Surgical and medical procedures) | 5
Aortic arteriosclerosis (Vascular disorders) | 1
Flushing (Vascular disorders) | 1
Haematoma (Vascular disorders) | 2
Hypertension (Vascular disorders) | 15
Hypotension (Vascular disorders) | 1
Varicose vein (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.